CLINICAL TRIAL: NCT02570282
Title: A Phase 2A, Single-Dose, Double-Blind Placebo-Controlled, 2-Way Crossover Study to Evaluate the Efficacy and Safety of SST-6007, a Topical Sildenafil Cream, Compared to Placebo in Women With Female Sexual Arousal Disorder
Brief Title: Study to Evaluate the Efficacy and Safety of SST-6007, a Topical Sildenafil Cream, Compared to Placebo in Women With Female Sexual Arousal Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Strategic Science & Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SST-6007-02-01
Record Dates: First submitted 2015-10-03; First posted 2015-10-07 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-01

CONDITIONS: Sexual Arousal Disorder
Keywords: Female
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil (Experimental): SST-6007 is a white to off-white cream containing 5% (w/w) sildenafil citrate
  Interventions: Drug: SST-6007
- Placebo (Placebo Comparator): Placebo IP will be the same as SST-6007 without the active ingredient, sildenafil citrate. It will be matched in appearance, smell, consistency, and color to SST-6007
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Approximately 50% of the cream is to be applied externally to the clitoris and labia minora and approximately 50% is to be applied intravaginally.
  Arms: Placebo
Drug: SST-6007 — SST-6007 is a white to off-white cream containing 5% (w/w) sildenafil citrate
  Arms: Sildenafil

SUMMARY:
This is a Phase 2, single center, single-dose, double-blind, placebo-controlled, 2-way crossover study to evaluate the safety and efficacy of SST-6007 in women with FSAD. A sufficient number of participants will be enrolled to yield 30 (approximately 15 pre-menopausal and 15 post-menopausal) participants to complete the SST-6007/Placebo Double-Blind, Dosing Phase of the study (Visit 2 and Visit 3).

DETAILED DESCRIPTION:
Participants will first complete a telephone screen (< 28 days prior to Visit 1, Medical Screening) and will be scheduled for Visit 1 if eligible. After consent is obtained, study participants will undergo Visit 1 at a local gynecology clinic to determine their eligibility for continued study participation.

If the participant meets all of the inclusion criteria and none of the exclusion criteria, they will be scheduled for Visit 2 and Visit 3 of the SST-6007/Placebo Double-Blind, Dosing Phase to be conducted at the Sexual Psychophysiology Laboratory at the University of Texas at Austin. Visit 2 must be within 5 (±2) days of Visit 1. One visit will evaluate the participant's response to SST-6007 and the other will evaluate the participant's response to placebo cream, using the VPP, the Arousometer, and neutral-erotic film presentations. The sequence of dosing will be randomly assigned (i.e., placebo cream then SST-6007 or SST-6007 then placebo cream) according to a computer-generated, randomization. There will be a 4-8 day washout period between Visits 2 and 3.

During each experimental session, physiological and subjective sexual arousal will be assessed simultaneously and continuously using the VPP and the Arousometer. Electrical activity of the heart will be assessed with an ECG. ECG data will be used to process the VPA data. Immediately following completion of each erotic film, subjective sexual arousal, subjective perception of genital arousal, and positive and negative affect will be evaluated using a self-report 7-point Likert Scale (Film Scale) and the Positive and Negative Affect Schedule (PANAS).

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal women (surgically induced or natural) must meet 1 of the following criteria:

   * Surgical oophorectomy, partial hysterectomy, or full hysterectomy at least 1 year prior to screening (self-report).
   * No spontaneous menses >1 year (self-report).
2. Post-menopausal participants, who are not on any hormone replacement therapies (HRT), must have a serum follicle-stimulating hormone (FSH) lab result >40mIU/mL.
3. Women of childbearing potential must agree to continue using an appropriate form of birth control from Visit 1 through 7 days following the completion of Visit 3. Acceptable forms of birth control include the use of an IUD or hormonal therapy (oral, patch, etc.). Contraceptive foams/gels or condoms are not considered acceptable methods of birth control in this study. Participants must be on a stable dose for at least 6 months prior to Visit 1.
4. Participant has a body mass index (BMI) from 18 to 30 kg/m², inclusive.
5. Participant is heterosexual.
6. Participant has a normal electrocardiogram at Visit 1.
7. Participant is capable of understanding and complying with the protocol and agrees to sign the informed consent document.
8. Participant must agree to not use vaginal or vulvar lubricants, spermicides, creams or gels, contraceptive foams or vaginal douche products from Visit 1 until the completion of Visit 3 9 Participant agrees to not engage in strenuous, unaccustomed exercise within 6 hours of visit 2 or visit 3.

Exclusion Criteria:

1. Participant is nursing or pregnant (based on positive serum pregnancy test), or wishes to become pregnant during the study period.
2. Participant has any disorder or a history of any disorder that may prevent the successful completion of the study in the opinion of the Sub-Investigator.
3. Participant has used any topical hormone replacement therapy (HRT) applied locally to the genitals in the past three months. Oral and patch form of HRT are acceptable, as long as the participant reports being on a stable dose for at least 6 months prior to Visit 1.
4. Participant has a significant cardiovascular, hepatic, metabolic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, genitourinary, or psychiatric disease or other unstable medical condition that would contraindicate administration of study medication, interfere with study evaluation, limit study participation, or confound the interpretation of study results in the opinion of the Sub-Investigator.
5. Participant had an active ulcer or clinically significant bleeding disorder.
6. Participant has a history of myocardial infarction, stroke, or life-threatening arrhythmia within 6 months prior to Visit 1; or any history of coronary disease causing angina; or congestive heart failure requiring medical intervention.
7. Participant has retinitis pigmentosa or sickle cell anemia or related anemias, even if the participant feels clinically well at the time of Visit 1. Participants with retinitis pigmentosa will be identified by specifically asking whether they have the condition, if there are visual signs and symptoms of the condition (including questioning participants as to whether they have difficulty seeing at night or in low light, and if they have any visual field deficits that indicate a loss of peripheral or central vision), or if there is a family history.

8 Participant has a history of orthostatic hypotension or orthostatic hypotension which is present at Visit 1, defined as a drop in systolic blood pressure ≥ 20 mm Hg, a drop in diastolic blood pressure ≥ 10 mm Hg or experiencing lightheadedness or dizziness at 1 or 3 minutes after the change in position from supine to standing.

9. Participant has primary anorgasmia, vaginismus, or sexual aversion disorder.

10. Participant has dyspareunia.

11. Participant has type 1 or type 2 diabetes.

12. Participant has undergone major pelvic surgery that may have caused nerve damage, including, vulvectomy, colostomy, cystostomy, or serious bladder, rectal, or abdominal surgery; neurological impairment due to diabetes, stroke, pelvic nerve damage secondary to trauma, cancer treatments, myasthenia gravis, multiple sclerosis or spinal cord damage.

13. Participant has current and/or previous reported diagnoses of DSM-IV-TR axis I disorders including organic mental syndromes and disorders (e.g., schizophrenia, bipolar disorder, depression).

14. Participant has a history of cancer, other than basal cell carcinoma.

15. Participant has any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article in the opinion of the Sub-Investigator.

16. Participant has a history of non-arteritic ischemic optic neuropathy (NAION).

17. Participant has positive findings from the urine drug screen (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, and opiates).

18. Participant has positive serologic findings for sexually transmitted infection (syphilis, gonorrhea, chlamydia), human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies.

19. Participant has moderate to severe current vaginitis, a vaginal infection including bacterial vaginosis or a yeast infection. The diagnosis of yeast infections should be made by the Sub-Investigator based on the physical and gynecological exams; the objective is to exclude women that are symptomatic. If the woman is not complaining of symptoms but the Sub-Investigator observes discharge, than the vaginal wet mount test should also be performed to confirm a diagnosis of yeast infection.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Participant-reported levels of subjective sexual arousal measured continuously by the Arousometer | 1 hour
  Measured on a 1-7 numeric scale evey 2 seconds
Physiological genital response in women with FSAD assessed using the vaginal photoplethysmograph (VPP) | 1 hour
  Measured on a 1-10 scale by electrical impulse 6 times a second

SECONDARY OUTCOMES:
Adverse events and vital signs | 21 days
  Adverse events and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Meston, PhD, Principal Investigator — University of Texas
Locations (1):
- The Sexual Psychophysiology Laboratory, Austin, Texas, United States